CLINICAL TRIAL: NCT04128787
Title: A Phase 1, Open-Label Study to Compare the Relative Bioavailability of Two AG-881 Formulations and to Evaluate the Effect of Food and Multiple-Dose Omeprazole on the Pharmacokinetics of a Single Dose of AG-881 in Healthy Adult Subjects
Brief Title: A Study to Compare the Relative Bioavailability of Two AG-881 Formulations and Evaluate the Effect of Food and Omeprazole on the Pharmacokinetics of AG-881
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG881-C-007
Record Dates: First submitted 2019-10-04; First posted 2019-10-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability Study; Pharmacokinetic study; AG-881
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Sequence ABCD (Experimental): Participants will receive Treatment A (AG-881 Formulation 1, 50 mg, tablet orally, under fasted condition once on Day 1 of Period 1) followed by Treatment B (AG-881 Formulation 2, 50 mg, tablet orally, under fasted condition once on Day 1 of Period 2) followed by Treatment C (AG-881 Formulation 2, 50 mg, tablet, orally, under fed condition once on Day 1 of Period 3) followed by Treatment D (omeprazole 40 mg capsule, orally, once daily on Days 1 to 4 and AG-881 Formulation 2, 50 mg, tablet, orally, under fasted condition, once on Day 4 of Period 4). Each period will be separated by a Washout Period of 21 days.
  Interventions: Drug: AG881 Formulation 1; Drug: AG881 Formulation 2; Drug: Omeprazole
- Treatment Sequence BCAD (Experimental): Participants will receive Treatment B in Period 1 followed by Treatment C in Period 2 then Treatment A in Period 3 followed by Treatment D in Period 4. Each period will be separated by a Washout Period of 21 days.
  Interventions: Drug: AG881 Formulation 1; Drug: AG881 Formulation 2; Drug: Omeprazole
- Treatment Sequence CABD (Experimental): Participants will receive Treatment C in Period 1 followed by Treatment A in Period 2 then Treatment B in Period 3 followed by Treatment D in Period 4. Each period will be separated by a Washout Period of 21 days.
  Interventions: Drug: AG881 Formulation 1; Drug: AG881 Formulation 2; Drug: Omeprazole

INTERVENTIONS:
Drug: AG881 Formulation 1 — AG881 uncoated tablets
Drug: AG881 Formulation 2 — AG881 film-coated tablets
Drug: Omeprazole — Omeprazole capsules

SUMMARY:
The purpose of this study is to compare the single-dose pharmacokinetics (PK) of two formulations (Formulation 1 and Formulation 2) of AG-881 and to examine the effect of food and multiple-dose omeprazole on the single-dose PK of AG-881 Formulation 2 in healthy adult participants. This study will also assess the safety and tolerability of single-dose AG-881 (Formulation 1 and 2) alone and of AG-881 Formulation 2 when administered with and without food and when coadministered with omeprazole in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (WONCBP) participants, 18-55 years of age, inclusive, at Screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECG, as deemed by the Investigator or designee. Liver function tests (serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and bilirubin [total and direct]) must be ≤ the upper limit of normal (ULN).
5. Female participants must be of non-childbearing potential defined as a female who has undergone one of the following sterilization procedures at least 6 months prior to the first dosing: hysteroscopic sterilization; bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy or is postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. A non-vasectomized, male participants must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing of study drug. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non-vasectomized male).
7. If a male participants, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Participant is mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or pose an additional risk to the participant (e.g., history or presence of rashes) by their participation in the study.
4. History of stomach or intestinal surgery that would potentially alter absorption/secretion; or any major surgical procedure within the previous 3 months prior to Screening.
5. History of severe and/or uncontrolled ventricular arrhythmias, or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome).
6. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
7. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
8. Any positive responses on the C-SSRS.
9. Female participants of childbearing potential.
10. Female participants with a positive pregnancy test or who are lactating.
11. Positive urine drug or alcohol results at Screening or first check-in.
12. Positive results at Screening for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.
13. QT interval Fridericia's formula (QTcF) interval is >450 msec, or QRS interval >110 msec, or PR interval >220 msec, or participants who have ECG findings deemed abnormal with clinical significance by the Investigator or designee at Screening.
14. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at Screening.
15. Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at Screening.
16. Estimated creatinine clearance <90 mL/min at Screening.
17. Unable to refrain from or anticipates the use of: Any drug, including prescription and non-prescription medications, herbal remedies, and vitamin supplements, beginning 14 days prior to the first dosing and throughout the study. After first dosing, ibuprofen (1.2 g per 24 hour) may be administered at the discretion of Investigator or designee. Hormone replacement therapy will not be allowed; any drugs known to be strong inducers of CYP3A, CYP2C9, or CYP2C19 enzymes including St. John's Wort and/or, gastric acid reducing agents (e.g., proton-pump inhibitors [with the exception of omeprazole administered as part of the study schedule], H2-receptor antagonists, antacids) for 28 days, or drugs that can prolong the QT interval for 21 days, prior to the first dosing and throughout the study. Appropriate sources (e.g., Flockhart TableTM) will be consulted to confirm lack of PK/Pharmacodynamic (PD) interaction with study drug.
18. Refuses to abstain from alcohol from 48 hours prior to the first dosing and throughout the study.
19. Refuses to abstain from grapefruit-containing foods or beverages or Seville orange containing foods or beverages from 14 days prior to the first dosing and throughout the study.
20. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
21. Any allergy or intolerance to food substances which will be provided on the study.
22. Is lactose intolerant.
23. Donation of blood or significant blood loss within 56 days prior to the first dose.
24. Plasma donation within 7 days prior to the first dose.
25. Receipt of blood or blood products within 2 months prior to the first dose.
26. Participation in another clinical study within 30 days prior to the first dose. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to the Last Observed Non-Zero Concentration (AUC0-t) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Concentration-Time Curve From Time 0 to the Last Observed Non-Zero Concentration (AUC0-t) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Maximum Observed Concentration (Cmax) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Maximum Observed Concentration (Cmax) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Concentration-Time Curve, From Time 0 to 504 Hours Postdose (AUC0-504) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Concentration-Time Curve, From Time 0 to 504 Hours Postdose (AUC0-504) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Terminal Elimination Half-life (t½) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Terminal Elimination Half-life (t½) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Time Delay Between Drug Administration and the Onset of Absorption (tlag) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Time Delay Between Drug Administration and the Onset of Absorption (tlag) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Time to Reach Maximum Observed Concentration (Tmax) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Time to Reach Maximum Observed Concentration (Tmax) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Volume of Distribution After Oral (Extravascular) Administration (Vd/F) of AG-881 Formulation 1 without Food | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Volume of Distribution After Oral (Extravascular) Administration (Vd/F) of AG-881 Formulation 2 with Food, without Food and when Co-administered with Omeprazole | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881

SECONDARY OUTCOMES:
Number of Participants with Abnormalities in Triplicate 12-lead Electrocardiograms (ECGs) | Up to 21 days in Period 1, 2, 3 (Each period is 21 days); up to 25 days in Period 4 (Period 4 is 25 days)
Number of Participants with Abnormalities in Vital Sign Measurements | Up to 21 days in Period 1, 2, 3 (Each period is 21 days); up to 25 days in Period 4 (Period 4 is 25 days)
  Vital sign measurements will include body temperature, respiratory rate, blood pressure, and heart rate.
Columbia-suicide Severity Rating Scale (C-SSRS) Score | Up to 21 days in Period 1, 2, 3 (Each period is 21 days); up to 25 days in Period 4 (Period 4 is 25 days)
  The C-SSRS is a questionnaire scale to detect emergent suicide symptoms (suicidal ideation or actual suicidal behavior) during the course of this study. Questions are either answered yes/no or are on a scale of 1 (low severity) to 5 (high severity).
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 21 days in Period 1, 2, 3 (Each period is 21 days); up to 25 days in Period 4 (Period 4 is 25 days)
  Clinical laboratory assessments will include hematology, serum chemistry, coagulation, and urinalysis.
Number of Participants with Adverse Events (AEs) | Up to 28 Days After Last Dose of Study Drug (Up to 91 days)'
  An AE is any untoward medical occurrence associated with the use of a drug, whether or not considered drug-related.
Number of Participants with Abnormalities in Physical Examinations | Up to 21 days in Period 1, 2, 3 (Each period is 21 days); up to 25 days in Period 4 (Period 4 is 25 days)
  Physical examination will include, examination of skin, neurological, respiratory, cardiovascular, and gastrointestinal systems.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No